CLINICAL TRIAL: NCT03475082
Title: Use of Modulating Frequency or Increasing Intensity to Overcome Analgesic Tolerance to Transcutaneous Electrical Nerve Stimulation (TENS) in Healthy Adults
Brief Title: Overcoming Analgesic Tolerance to TENS
Acronym: OCTTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen Sluka (Other)
Responsible Party: Sponsor-Investigator, Kathleen Sluka, PT, PhD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201203735
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial -double blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo TENS (Placebo Comparator): 30 minute TENS treatment where the stimulation ramps slowly to zero after 45 seconds. The lights/display on the unit are identical to the Active unit.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- High Frequency TENS (Active Comparator): 30 minute TENS treatment at 100 Hertz (HZ). Intensity set at a strong but comfortable setting and subject asked to increase intensity as tolerated every 5 minutes. Final stimulation intensity at end of Day 1 treatment used for the remainder of the treatment sessions for all 5 days.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Alternating frequency TENS (Active Comparator): 30 minute TENS treatment with a pre programed mode alternating from 4 Hz and 100 HZ. Intensity set at a strong but comfortable setting and subject asked to increase intensity as tolerated every 5 minutes. Final stimulation intensity at end of Day 1 treatment used for the remainder of the treatment sessions for all 5 days.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Modulated frequency TENS (Active Comparator): 30 minute TENS treatment at a pre programmed mode that ramps between 4 and 125 HZ over 12 seconds. Intensity set at a strong but comfortable setting and subject asked to increase intensity as tolerated every 5 minutes. Final stimulation intensity at end of Day 1 treatment used for the remainder of the treatment sessions for all 5 days.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- High frequency TENS - increasing intensity (Active Comparator): 30 minute TENS treatment at 100 HZ. Intensity set at initial strong but comfortable setting on day one as above, then subjects asked for possible increases in intensity every 5 minutes on all five days.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous electrical nerve stimulation (TENS) is utilized clinically by a variety of health care professionals for the reduction of pain. The mechanisms by which TENS produces analgesia or reduces pain are only recently being elucidated. TENS is a non-invasive modality that is inexpensive, safe and easy to use with relatively few contraindications. Frequency of stimulation is broadly classified as high frequency (>50Hz), low frequency (<10Hz) TENS. Intensity is determined by the response of the patient as either sensory level (low-intensity) TENS strong but comfortable. With sensory level TENS, the voltage (i.e. amplitude) is increased only until the patient feels a comfortable tingling (perceived with high frequency) or tapping (perceived with low frequency) sensation without motor contraction. With strong but comfortable TENS the intensity is increased to a strong but comfortable level which may include muscle contraction.
  Other Names: TENS; Electrical stimulation

SUMMARY:
The purpose of this study is to determine if changing the frequency or intensity of transcutaneous electrical nerve stimulation (TENS) can reduce the development of tolerance to TENS treatment.

DETAILED DESCRIPTION:
Healthy adults will come daily for 5 consecutive days to the testing room. Pressure pain thresholds (PPT) will be the outcome measure and will be used to measure the subject's pain threshold to deep mechanical pressure. Subjects will push a button to stop the PPT test when they first begin to feel a sensation of pain. The PPT test will be done before TENS application. The TENS unit will be applied based on random assignment to 1 of 5 treatment types and subjects will not be told which group they are assigned to. Those groups are: 1) placebo TENS, 2) high frequency TENS, 3) alternating frequency TENS, 4) modulated frequency TENS, or 5) high frequency TENS with increased intensity daily. The TENS unit will be applied for 30 minutes. After 20 minutes the PPT test will be completed a second time. This procedure will occur on all 5 consecutive days of testing. Data will be measured and recorded by an assessor blind to subject group. Blinding will be assessed at the end of testing on day 5.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 Years of Age (YOA)
* no current pain condition

Exclusion Criteria:

* Pregnancy
* Cardiac pacemaker
* Currently experiencing pain
* Abnormal sensation in dominant forearm
* History of seizures
* Prior TENS use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Pre TENS and post TENS at initial (day 1) and final (day 5) study visit
  Pressure pain thresholds (PPTs) change score measured in kilopascal (kPa) will be assessed on the forearm using a pressure algometer. The pressure algometer is mechanical pressure applied by the research assistant at a gradual rate by pushing the device against the skin. The device has a 1 cm2 pad that is in contact with the skin. The subject has a button that they push when the pressure first becomes painful (threshold)which stops the test and the pressure amount is recorded by the research assistant. This is the amount of pressured in kPa that is required to cause a subjective pain of 1/10 on a scale of 0 (no Pain) to 10 (Maximum Pain) rating by the subject. The change score from day 1 to Day 5 is the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Sluka, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandran P, Sluka KA. Development of opioid tolerance with repeated transcutaneous electrical nerve stimulation administration. Pain. 2003 Mar;102(1-2):195-201. doi: 10.1016/s0304-3959(02)00381-0. PMID 12620611
- [Background] Desantana JM, Santana-Filho VJ, Sluka KA. Modulation between high- and low-frequency transcutaneous electric nerve stimulation delays the development of analgesic tolerance in arthritic rats. Arch Phys Med Rehabil. 2008 Apr;89(4):754-60. doi: 10.1016/j.apmr.2007.11.027. PMID 18374009
- [Background] Liebano RE, Rakel B, Vance CGT, Walsh DM, Sluka KA. An investigation of the development of analgesic tolerance to TENS in humans. Pain. 2011 Feb;152(2):335-342. doi: 10.1016/j.pain.2010.10.040. Epub 2010 Dec 8. PMID 21144659